CLINICAL TRIAL: NCT00096980
Title: An Open Label, Randomized, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneously Administered Efalizumab Used in Combination With Topical Psoriasis Therapies for Prolonged Maintenance Treatment
Brief Title: A Study to Evaluate Raptiva in Combination With Topical Psoriasis Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ACD2243g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva (efalizumab)

SUMMARY:
This study is an open label, randomized, multicenter study designed to compare the efficacy of 12 weeks of subcutaneously administered efalizumab (monotherapy) with that of combination therapy (Efalizumab and a topical corticosteroid ointment) in subjects with moderate to severe plaque psoriasis who are candidates for systemic therapy. The study will also evaluate the safety and tolerability of 30 months of continuous efalizumab treatment in those subjects who derive benefit from the initial 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of plaque psoriasis for >=6 months
* A minimum Psoriasis Area and Severity Index (PASI) score of 12.0 at screening
* Plaque psoriasis covering >=10% of total Body Surface Area (BSA)
* In the opinion of the investigator, candidate for systemic therapy for psoriasis who has not been previously treated (naive to systemic treatment) or who has received prior systemic therapy for psoriasis (e.g., PUVA, cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil [MMF], thioguanine, hydroxyurea, sirolimus, azathioprine, 6 MP, etanercept)
* 18 to 70 years old

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* Clinically significant psoriasis flare during the 3 months prior to enrollment
* Pregnancy or lactation
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for hepatitis B or C virus
* Seropositivity for human immunodeficiency virus (HIV)
* History of active tuberculosis (TB) or currently undergoing treatment for TB
* Presence or history of malignancy within the past 5 years, including lymphoproliferative disorders
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Hospital admission for cardiovascular or pulmonary disease within the last year
* History of substance abuse within the last 5 years
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or fusion proteins, which contain an immunoglobulin (Ig) Fc region (e.g., etanercept, LFA3TIP)
* History of severe allergic reactions to or intolerance of topical corticosteroid therapies
* Previous treatment with efalizumab
* History of treatment with lymphocyte-depleting monoclonal antibodies or immunoadhesion molecules (e.g., anti-CD4, CTLA4-Ig, LFA3TIP)
* WBC count <4000/uL or >14,000/uL
* Hepatic enzymes >=3 times the upper limit of normal
* Creatinine >=2 times the upper limit of normal
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug
* Any medical or other condition that, in the judgment of the investigator, would significantly interfere with the subject's ability to comply with the provisions of this protocol
* Topical therapy for psoriasis
* Systemic therapy for psoriasis
* Systemic immunosuppressive drugs
* Tanning beds, booths, or home UV light sources
* Live virus or bacteria vaccine
* Other vaccines or allergy desensitization injections
* Other experimental drugs or treatments
* Nonsteroidal anti inflammatory drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-02; Study Completion 2004-05 (Actual)

REFERENCES:
- [Derived] Lamerson C, Stevens G, Sax K. Treatment of nail psoriasis with efalizumab: a preliminary study. Cutis. 2008 Sep;82(3):217-20. PMID 18856162